CLINICAL TRIAL: NCT06845124
Title: ICONICplus - Randomized, Double-blind, Placebo-controlled Trial to Investigate the Effects of Cannabidiol Plus Naltrexone on Cue-Induced Alcohol Craving in Alcohol Dependence
Brief Title: A Trial to Investigate the Effects of Cannabidiol Plus Naltrexone on Alcohol Craving in Patients With Alcohol Dependence
Acronym: ICONICplus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Heidelberg University - Institute of Medical Biometry (IMBI) (Unknown); Heidelberg University - Coordination Centre for Clinical Trials (KKS) of Heidelberg University (Unknown); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIMH ICONICplus 25; 2024-518164-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Addiction; Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Cannabidiol; Naltrexone; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cannabidiol (800mg) + Naltrexone (Experimental): All patients will receive 50mg Naltrexone daily (NTX, oral tablet) in the course of standard in-patient treatment. In the experimental group of trial arm 1, patients will receive a dose of 800mg Cannabidiol (CBD) daily over the course of 14 days during in-patient treatment.
  Interventions: Drug: Cannabidiol capsules; Drug: Naltrexone (drug)
- Cannabidiol (1200mg) + Naltrexone (Experimental): All patients will receive 50mg Naltrexone daily (NTX, oral tablet) in the course of standard in-patient treatment. In the experimental group of trial arm 2, patients will receive a dose of 1200mg Cannabidiol (CBD) daily over the course of 14 days during in-patient treatment.
  Interventions: Drug: Cannabidiol capsules; Drug: Naltrexone (drug)
- Placebo + Naltrexone (Active Comparator): All patients will receive 50mg Naltrexone daily (NTX, oral tablet) in the course of standard in-patient treatment. In the comparator group of trial arm 3, patients will receive placebo capsules daily over the course of 14 days during in-patient treatment.
  Interventions: Drug: Naltrexone (drug); Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol capsules — 800mg (trial arm 1) or 1200mg (trial arm 2) Cannabidiol capsules will be administered daily over the course of 14 days.
  Arms: Cannabidiol (1200mg) + Naltrexone; Cannabidiol (800mg) + Naltrexone
Drug: Naltrexone (drug) — All participants will receive 50mg Naltrexone daily as oral tablet throughout the study.
Drug: Placebo — Placebo capsules matching the cannabidiol capsules will be administered daily.
  Arms: Placebo + Naltrexone

SUMMARY:
Alcohol addiction (AD) is a chronic relapsing disorder with currently limited pharmacological treatment options. Alcohol craving, a hallmark symptom of AD that drives relapse in patients, is only insufficiently treated by existing medication. One promising new compound for the treatment of alcohol craving in AD is Cannabidiol (CBD), which showed beneficial effects on alcohol craving in preliminary clinical studies. Additionally, CBD seems to be a particularly promising candidate for enhancing the effects of established medication, specifically Naltrexone (NTX), an opioid-antagonist, which is approved for AD treatment, due to the synergistic effects of the combination of Cannabidiol plus Naltrexone on alcohol consumption that were shown by preclinical studies. The proposed three-armed, 1:1:1 randomized, double-blind, placebo-controlled parallel group, multicentric phase II trial seeks to test the putative synergistic effects of combined CBD (800mg) + oral NTX (50mg) against CBD (1200mg) + oral NTX (50mg) against Placebo + oral NTX (50mg) on alcohol craving (primary outcome) in male and female patients with AD that suffer from high alcohol craving. The trial seeks to test the effects of the innovative combination of CBD plus NTX against Placebo plus NTX on alcohol craving over a 14-day treatment period, which is embedded in a standardized addiction treatment program according to current treatment guidelines, in order to estimate the added value of treatment with CBD on alcohol craving. Quality of life and neurobiological and biochemical markers for craving will serve as secondary outcomes, because they show strong associations to treatment outcome and relapse risk. Collection and analysis of follow-up data (28 days, 42 days, 105 days, 196 days) will be performed to determine whether treatment effects relate to patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Patients meeting the diagnosis of an alcohol dependence according to the ICD-10
* Patients reporting alcohol craving as symptom of AD according to the ICD10 symptom definition
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrollment in the study)
* Consent to random assignment
* For women with childbearing potential (WOCBP) and males with partners with CBP, use of a highly effective birth control method until one month after last IMP administration (see Appendix 1) and negative pregnancy test

Exclusion Criteria:

* Current psychotic or bipolar disorder or current severe depressive episode with suicidal ideations
* Current treatment with any of the following substances: Any investigational medicinal product, Opioid-containing Analgesics, Anti-obesity drugs, Anticonvulsants, Opioid-containing Antidiarrheal Agents, Antineoplastics, Antipsychotics (exception: episodic use of melperone, prothipendyl, pipamperone, promethazine and quetiapine are allowed), Antidepressants (exception: allowed, when being taken in stable dose for a minimum of 14 days prior to enrolment and/or doxepine in low doses [max. 75mg daily]), Opioid-containing Cough/cold agents, Systemical Steroids, Other anti-craving (e.g. Acamprosate) or aversive medication (e.g. disulfiram), THC- or CBD-containing medication, Antiretroviral medication (e.g., Efavirenz), Xanthines (e.g., Theophylline), General anesthetics (e.g., propofol), Hypericum perforatum, Antibiotics (e.g., Rifampin, Clarithromycin, Erythromycin)
* Positive drug screening (amphetamines/ecstasy, opiates, cocaine, barbiturates)
* Pregnancy, lactation or breastfeeding
* Current severe somatic comorbidities: severe liver cirrhosis [CHILD B or C] or epilepsy determined by medical history
* Patients with elevated transaminase levels (AST or ALT) above three times the upper limit normal (ULN) value with elevated bilirubin levels above twice the ULN value
* History of hypersensitivity to the investigational medicinal product CBD and/or Naltrexone (trade names: Adepend, Naltrexon-Hcl neuraxpharm, Naltrexonhydrochlorid Accord) or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product CBD and/or Naltrexone
* Participation in other clinical trials or observation period of competing clinical trials, respectively.
* Acute suicidal tendency or acute endangerment of self and others

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Obsessive Compulsive Drinking Scale (OCDS-G) | The difference of alcohol craving between baseline (visit 2) and 14 days after the first treatment visit (visit 5) will serve as primary endpoint.
  The alcohol craving will be assessed at separate time points before and after Cannabidiol administration using the Obsessive Compulsive Drinking Scale.
  The Obsessive Compulsive Drinking Scale consists of 14 items, each rated on a 5-point Likert scale (0-4), resulting in scores from 0 to 40, with higher scores indicating higher craving.

SECONDARY OUTCOMES:
Obsessive Compulsive Drinking Scale (OCDS-G) | Differences from baseline (visit 2, day -2) of Obsessive Compulsive Drinking Scale craving scores to visits 4 (day 7, i.e., 7 days after the first treatment visit) and during follow up visits 6 (day 28), 7 (day 42), 8 (day 105), 9 (day 196)
  The alcohol craving will be assessed at separate time points before and after Cannabidiol administration using the Obsessive Compulsive Drinking Scale.
  The Obsessive Compulsive Drinking Scale consists of 14 items, each rated on a 5-point Likert scale (0-4), resulting in scores from 0 to 40, with higher scores indicating higher craving.
Subjective quality of life index | Differences from baseline (visit 2, day -2) of Quality of life (WHO-QOL-BREF scores) to end of treatment (visit 5, day 14) and follow up visits 6 (day 28), 7 (day 42), 8 (day 105), 9 (day 196).
  Quality of life will be assessed using the World Health Organization Quality of life questionnaire (WHO-QOL-BREF) scores at separate time points before and after Cannabidiol administration. The World Health Organization Quality of life questionnaire is an instrument that can assess patients' global health status independently of disease across 4 health domains and consists of 26 items rated on a 5-point Likert scale (1-5). To calculate the score, items 3, 4, 26 have to be inverted. Scores for each domain (Physical Health, Psychological Health, Social Relationships, Environment) are calculated, that range from 4 to 20. Higher scores indicate better quality of life, with the overall score reflecting a person's general well-being.
Beck Depression Inventory (BDI-II) | Difference from baseline (visit 2, day -2) of depressive symptoms to end of treatment (visit 5, day 14)
  The depressive symptoms will be assessed at separate time points before and after Cannabidiol administration using the Beck Depression Inventory (BDI-II). The Beck Depression Inventory (BDI-II) is a 21-item self-rating inventory that measures characteristic attitudes and symptoms of depression. Each Item is rated on a 4-point Likert scale (0-3). The total score ranges from 0 to 63, with higher scores indicating more severe depressive symptoms.
State Trait Anxiety Inventory (STAI) | Difference from baseline (visit 2, day -2) of depressive symptoms to end of treatment (visit 5, day 14)
  The state and trait anxiety will be assessed at separate time points before and after Cannabidiol administration using the State Trait Anxiety Inventory. The State Trait Anxiety Inventory (STAI) is a 20-item self-report questionnaire that assesses state anxiety and trait anxiety via two subscales: the State Anxiety Scale (STAI-S) and the Trait Anxiety Scale (STAI-T), each consisting of 20 items. Each item is rated on a 4-point Likert scale (1-4). A sumscore has to be calculated for each subscale, ranging from 20 to 80 each, with higher scores indicating higher levels of anxiety.
Patient reported outcomes (PRO) | On visit 3 (day 1 of treatment), visit 4 (day 7 of treatment), visit 5 (day 14, end of treatment) and during follow up visits 6 (day 28), 7 (day 42), 8 (day 105), 9 (day 196)
  The patient reported outcomes will be assessed at separate time points before and after Cannabidiol administration using a set of items assessing effects of the treatment as well as treatment burden on a five-point Likert scale (0 to 4) with higher values indicating more positive effects.
CBD plasma levels | On visit 3 (day 1 of treatment) and visit 5 (day 14, end of treatment)
  The CBD plasma levels will be determined at separate time points before and after Cannabidiol administration to detect effects of active intervention on blood plasma levels. (Only participants enrolled at CIMH study site).
Adverse Events (AEs) and Serious Adverse Events (SAEs) | On visit 3 (day 1 of treatment), visit 4 (day 7 of treatment), visit 5 (day 14, end of treatment) and during follow up visits 6 (day 28), 7 (day 42), 8 (day 105), 9 (day 196)
  Rate of adverse events and serious adverse events.
Time to relapse | On visit 5 (day 14, end of treatment) and during follow up visits 6 (day 28), 7 (day 42), 8 (day 105), 9 (day 196)
  Time from baseline (visit 2, day -2) to relapse to alcohol use (i.e. any alcohol use) (in days), assessed using the Form-90 semi-structured interview (Timeline Follow Back).
Cumulative alcohol consumption during the follow-up period | On visit 5 (day 14, end of treatment) and during follow up visits 6 (day 28), 7 (day 42), 8 (day 105), 9 (day 196)
  Cumulative alcohol consumption (in grams alcohol) during the follow-up period of 182 days (+/- 7 days), assessed using the Form-90 semi-structured interview (Timeline Follow Back).
Percent heavy drinking days during the follow-up period | On visit 5 (day 14, end of treatment) and during follow up visits 6 (day 28), 7 (day 42), 8 (day 105), 9 (day 196)
  Percent heavy drinking days during the follow-up period of 182 days (+/- 7 days), assessed using the Form-90 semi-structured interview (Timeline Follow Back).
Average weekly alcohol consumption during the follow-up period | Every 7 days during the follow-up period of 182 days (+/- 7 days), starting after visit 5, i.e., end of treatment (day 14) and continuing until visit 9, i.e., end of follow up (day 196)
  Average weekly alcohol consumption assessed via smartphone-based e-diary every 7 days during the follow-up period of 182 days (+/- 7 days) (optional, only for patients that agree to use the study-specific app).
Maximum weekly craving during the follow-up period | Every 7 days during the follow-up period of 182 days (+/- 7 days), starting after visit 5, i.e., end of treatment (day 14) and continuing until visit 9, i.e., end of follow up (day 196)
  Maximum weekly craving assessed via smartphone-based e-diary every 7 days during the follow-up period of 182 days (+/- 7 days) (optional, only for patients that agree to use the study-specific app).
Neural Brain Activation during functional magnetic resonance imaging | Differences from baseline (visit 2, day -2) to visit 5 (day 14, end of treatment)
  Differences from baseline of neural brain activation to visit 5, measured using the blood oxygenated level dependent (BOLD) response, during presentation of alcohol cues, during the presentation of natural reward cues, during inhibition of motor responses, during presentation of emotional faces and neutral shapes and functional connectivity during resting state (only for patients enrolled at CIMH study site).
Alcohol Craving during functional magnetic resonance imaging | Differences from baseline (visit 2, day -2) to visit 5 (day 14, end of treatment)
  Differences from baseline of alcohol craving (visual analogue scale) during the functional magnetic resonance imaging (fMRI) to visit 5 (only for patients enrolled at CIMH study site).
Response Times during functional magnetic resonance imaging | Differences from baseline (visit 2, day -2) to visit 5 (day 14, end of treatment)
  Differences in response times (i.e., time taken to respond) during functional magnetic resonance imaging (fMRI) from baseline to visit 5 (only for patients enrolled at CIMH study site).
Rates of Errors during functional magnetic resonance imaging | Differences from baseline (visit 2, day -2) to visit 5 (day 14, end of treatment)
  Differences in rates of errors during functional magnetic resonance imaging (fMRI) from baseline to visit 5 (only for patients enrolled at CIMH study site)
Rates of Correct Responses during functional magnetic resonance imaging | Differences from baseline (visit 2, day -2) to visit 5 (day 14, end of treatment)
  Differences in rates of correct responses during functional magnetic resonance imaging (fMRI) from baseline to visit 5 (only for patients enrolled at CIMH study site)
Omission Rates during functional magnetic resonance imaging | Differences from baseline (visit 2, day -2) to visit 5 (day 14, end of treatment)
  Differences in omission rates (i.e., rate of failure to respond when a response is expected) during functional magnetic resonance imaging (fMRI) from baseline to visit 5 (only for patients enrolled at CIMH study site)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Bach, Prof. Dr. Dr., Study Director — Central Institute of Mental Health, Mannheim
Locations (2):
- Germany (2):
  - Psychiatric Centre North Baden (PZN), Wiesloch, Baden-Wurttemberg
  - Central Institute of Mental Health, Mannheim

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified data will be shared, specifically individual participant data that underlie the results of the trial (i.e. primary outcome data [OCDS-G scores]) will be made available with a respective data dictionary. Secondary Outcome data (e.g. fMRI data) will be made available on aggregated group level (e.g. for the purpose of meta-analyses). Related documents, specifically the study protocol, statistical analysis plan and analytic code will be shared in open-access online repositories. Aggregated data will be made available to publicly accessible repositories (Neurosynth.org), e.g. for the purpose of meta-analyses.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available upon publication of the results until 3 years after that.
Access Criteria: Individual data will be shared with researchers who provide a methodologically sound proposal (sent to the Principal Investigator/Study Chair of the Trial).

REFERENCES:
- [Derived] Vetter S, Weinberg J, Thomas BC, Kirchner M, Thalmann P, Klose C, Pfisterer M, Kolsch T, Oesterle S, Vollstaedt-Klein S, Koopmann A, Lenz B, Kiefer F, Link T, Bach P. Investigation of the combined effects of cannabidiol plus naltrexone on alcohol craving in alcohol dependence: study protocol of a phase II randomised, double-blind, placebo-controlled, parallel-group trial - ICONICplus Trial. BMJ Open. 2025 Aug 12;15(8):e106348. doi: 10.1136/bmjopen-2025-106348. PMID 40803733